CLINICAL TRIAL: NCT05329779
Title: Using Allopregnanolone to Probe Behavioral and Neurobiological Mechanisms That Underlie Depression in Women During the Perimenopause
Brief Title: Study on Allopregnanolone and Depression in Perimenopausal Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hadine Joffe, MD MSc, Study Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P003137
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — brexanolone; Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- brexanolone (Experimental): Participants will receive a continuous 60-hr intravenous infusion of brexanolone
  Interventions: Drug: brexanolone
- placebo (Placebo Comparator): Participants will receive a continuous 60-hr infusion of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: brexanolone — Brexanolone is a derivative of allopregnanolone, which is FDA-approved to treat postpartum depression.
  Other Names: Zulresso; allopregnanolone
  Arms: brexanolone
Drug: placebo — The placebo is a 0.45% sodium chloride infusion.
  Arms: placebo

SUMMARY:
This study aims to identify how the progesterone metabolite allopregnanolone affects behavior and neurobiology that may underlie perimenopausal depression.

DETAILED DESCRIPTION:
Midlife women are burdened with depression risk that is at least partly attributed to changing reproductive steroid dynamics across a prolonged reproductive transition. The investigators hypothesize that declining endogenous allopregnanolone (ALLO) levels across the menopause transition underlies perimenopausal depression. This mechanistic trial aims to amplify the contrast between lower endogenous ALLO levels in perimenopausal women and higher levels experimentally induced by exogenous ALLO. This will be achieved by using the exogenous ALLO treatment, brexanolone, which is FDA-approved to treat depression in postpartum patients, in a randomized, double-blind, parallel-arm, placebo-controlled trial. By manipulating ALLO levels together with key measurement of depression domains, this study harnesses the endocrine biology of perimenopause to explicate behavioral and neurobiological mechanisms underlying depression in perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy perimenopausal women ages 40 to 60 years
* Depressive symptoms
* Able to read Arabic numerals and perform simple arithmetic
* Able to provide written informed consent

Exclusion Criteria:

* Use of medications to treat depression
* Systemic hormone therapy
* Contraindicated medications with brexanolone
* Other psychiatric illnesses that are considered to be primary
* Current suicidal ideation
* Active substance use disorders
* Unstable medical conditions
* Obstructive sleep apnea or other primary sleep disorders
* Abnormal hepatic and renal function
* Known allergy to progesterone, exogenous allopregnanolone, or brexanolone
* History of head injury resulting in loss of consciousness > 20 min
* Inability to comply with barrier contraceptive methods
* Known intellectual disability
* Investigator judgement that study participation constitutes substantial risk given medical or psychiatric condition
* Current or recent participation in clinical trial expected to interfere with risk of or interpretation of study data
* Inability to comply with study procedures

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brexanolone | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Results are not posted due to potential risk to confidentiality given low enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexanolone | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Within-person Change in Score on the Ruminative Responses Scale
Description: The Ruminative Responses Scale (RRS) comprises 22 items which ask how frequently the participant thinks certain statements when they feel depressed. Each item is scored from 1-4. Total scores range from 22-88 with higher scores indicating more severe rumination.
Time Frame: Baseline to 4 days
Population: Results are not posted due to potential risk to confidentiality given low enrollment.
Arm/Group | Brexanolone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 30 days
Description: Adverse events are not posted due to potential risk to confidentiality given low enrollment.
Arm/Group | Brexanolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to operational feasibility. The decision to terminate the study was not related to any new or emerging safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05329779/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05329779/ICF_001.pdf